CLINICAL TRIAL: NCT01636635
Title: Effect of Age and Weight Loss on Obesity-related Inflammation and Iron Homeostasis in Women
Brief Title: Effect of Age and Weight Loss on Inflammation and Iron Homeostasis
Acronym: HEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Simin Meydani, Simin Meydani, DVM, PhD, Tufts University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2765
Record Dates: First submitted 2012-01-26; First posted 2012-07-10 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Obesity; Aging
MeSH Terms: conditions — Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Young (18-45 years) (Active Comparator): Obese young women (18-45y) undergoing calorie restriction.
  Interventions: Other: Calorie Restriction
- Older (>60 years) (Experimental): Obese older women (>60y) undergoing calorie restriction.
  Interventions: Other: Calorie Restriction

INTERVENTIONS:
Other: Calorie Restriction — Intervention consists of a calorically restricted diet regime designed and administered at the Weight and Wellness Center at Tufts University

SUMMARY:
The purpose of this study is to evaluate the effect of aging and weight loss on iron status and immune response in obese women. Iron deficiency and immune impairment are two of the numerous complications of obesity. The central hypothesis is that obesity-induced inflammation causes lower iron status through decreased iron absorption and availability in young and older obese women. Furthermore, the investigators hypothesize that this can be corrected with weight loss in both young and older obese women.

DETAILED DESCRIPTION:
Obese individuals have chronic inflammation, higher risk of iron deficiency, and impaired immune response. These are conditions seen also with aging, but it is unknown to what extent they may be further impacted by obesity in the elderly. With this study the investigators aim to establish the mechanism by which weight loss may reduce inflammation and enhance iron status in young and older obese adults through the peptide hormone hepcidin, which regulates iron homeostasis. The investigators also aim to identify a possible link between iron homeostasis and immune response through hepcidin, which has been implicated in T cell mediated immunity. The investigators hypothesize that obesity-induced inflammation causes dysregulation of hepcidin expression leading to lower iron status through decreased iron absorption and availability in young and older adults. Furthermore, the investigators hypothesize that hepcidin dysregulation, and thus iron status can be mitigated with weight loss in both young and older obese adults. This hypothesis will be tested in obese young and older women undergoing weight loss through calorie restriction. Change in iron status, inflammation, and hepcidin will be determined before and after weight loss. Further, the impact of inflammatory environment of obesity on peripheral blood mononuclear cell hepcidin, ferroportin, intracellular iron, and T cell function in young and older adults will be determined. This study will address two important public health problems, i.e. obesity and iron deficiency and will be an important step toward the identification of strategies to enhance health of obese young and older adults.

ELIGIBILITY:
Inclusion Criteria:

* Enrolling patients in the Weight and Wellness Center (WWC) at Tufts Medical Center, part of their Tufts Employees, low calorie diet (LCD) or pre-surgical low calorie diet (PS-LCD) program, or enrolling at WWC as individual patients.
* BMI in the range of 30 to 55 kg/m2.
* Either ages 18-45 or >60.

Exclusion Criteria:

* Pregnancy.
* Weight reduction greater than or equal to 3% in the past 3 months.
* Prior gastric restrictive surgery.
* Weight loss medications within the 4 weeks prior to screening.
* History of eating disorder.
* Renal disease (serum creatinine >2mg/dl).
* Hepatic disease, except for nonalcoholic steatohepatitis (NASH).
* Celiac disease, or any kind of intestinal malabsorption disorders.
* Gastrointestinal cancer.
* Hereditary hemochromatosis, or any blood disorders.
* Chronic infectious or inflammatory disease.
* Use of immunosuppressants.
* Severe iron deficiency anemia (hemoglobin<8 g/dl) or other conditions that would prevent them from discontinuing iron supplement use.
* Unwilling to discontinue iron supplement intake. The dietary plan recommended by the WWC will include daily intake of iron that meets the iron RDA for the subject's gender and age group, therefore discontinuing iron supplement will not be harmful for the participants. Intake of other supplements will not be an exclusion criteria, as long as it stays constant throughout the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in serum hepcidin | Baseline and 12-16 weeks
  The investigators will determine the change in hepcidin at baseline and after 12-16 weeks of calorie restriction.
Change in inflammation (CRP, IL-6) | Baseline and 12-16 weeks
  The investigators will determine the change in inflammation at baseline and after 12-16 weeks of calorie restriction.
Change in iron status | Baseline and 12-16 weeks
  The investigators will determine the change in iron status at baseline and after 12-16 weeks of calorie restriction.

SECONDARY OUTCOMES:
Change in PBMC intracellular iron content | Baseline and 12-16 weeks
Change in PBMC Hepcidin expression | Baseline and 12-16 weeks
Change in PBMC ferroportin expression | Baseline and 12-16 weeks
Change in PBMC subpopulations and proliferation | Baseline and 12-16 weeks
  After stimulation with ConA, PHA and anti-CD3/CD28

CONTACTS AND LOCATIONS:
Overall Officials: Simin N Meydani, DVM, PhD, Principal Investigator — Tufts University
Locations (1):
- JM USDA Human Nutrition Research Center on Aging, Boston, Massachusetts, United States